CLINICAL TRIAL: NCT01448772
Title: A Single-Dose, Replicate Crossover Design Comparative Bioavailability Study of Dronabinol Oral Solution 5 mg Versus Marinol Capsules 5 mg Under Fasted Conditions
Brief Title: Comparative Bioavailability of Dronabinol Oral Solution Versus Branded Capsule 5 mg Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: INSYS Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: INS-10-012
Record Dates: First submitted 2011-10-05; First posted 2011-10-07 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Bioavailability
Keywords: Dronabinol; fasting
MeSH Terms: conditions — Fasting | interventions — Dronabinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Marinol (Active Comparator)
  Interventions: Drug: Dronabinol Capsules, 5 mg
- oral solution (Experimental)
  Interventions: Drug: Dronabinol Oral Solution

INTERVENTIONS:
Drug: Dronabinol Capsules, 5 mg — Comparison of different routes of administration of a drug using the approved Abbott 5 mg capsule product under fasting conditions; two treatment periods with a washout period separating the study periods
  Arms: Marinol
Drug: Dronabinol Oral Solution — Comparison of different routes of administration of a drug using a proposed oral solution formulation under fasting conditions; two treatment periods with a washout period separating the study periods
  Arms: oral solution

SUMMARY:
This is a comparative study to assess bioavailability of a proposed alternate dosage form against the current FDA-approved branded product.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female healthy subjects between 18 and 55 years of age, inclusive.
2. Subjects must have a body mass index (BMI) within 19 and 29.9 kg/m2, inclusive and weigh a minimum of 50 kg (110 pounds).
3. Subjects must be in general good health as determined by medical history, physical examination, or laboratory evaluations conducted at the screening visit and upon admission to the clinic. Examination should include a thorough examination of oral cavity for any abnormal findings.
4. Subjects must be non-smokers, defined as not having used any tobacco products in the past six months. Negative results from a urine cotinine test conducted at Screening.
5. Subjects must be able to provide informed consent after risks and benefits have been explained, and be willing to comply with study procedures.
6. Female subjects of childbearing potential must not be pregnant or nursing; and must be surgically sterile; one year postmenopausal; or on hormonal contraceptive agent(s), diaphragm or condom with spermicidal foam or jelly, or IUD for at least three months prior to drug administration and agree to use the same method of contraception for at least one month after the last drug administration.
7. Negative urine pregnancy test at screening and prior to drug administration of each period.
8. Negative HIV 1, hepatitis C virus (HCV) antibody, hepatitis B surface antigen within 30 days prior to the start of the study.
9. Negative results from screening for drugs of abuse at Screening and Day-1 (check-in) prior to drug administration during all study periods.

Exclusion Criteria:

1. Known hypersensitivity or allergy to dronabinol, Marinol, marijuana, hashish, or sesame oil.
2. Have participated in an investigational trial within 30 days or six half-lives of the test drug's biologic activity, whichever is longer, before the time of first study dose in this study.
3. Presence of visible signs of an infection, mucositis, cold sores, lesions, local irritation, periodontal disease of the oral cavity or any abnormal finding in the oral cavity. In addition, evidence of piercings of the tongue, lip, or anywhere in the oral cavity or a history of oral cavity piercings.
4. Have donated or received blood or blood products within 30 days prior to the first study dose.
5. Have received any prescription drug (excluding hormonal contraceptives) within 14 days of study drug administration, over-the-counter drugs within seven days of study drug administration, and/or vitamins or herbal supplements within three days of study drug administration.
6. Significant bradycardia or tachycardia defined as having a resting heart rate <45 bpm or >100 bpm, respectively.
7. Clinical evidence of either hypotension (defined as systolic blood pressure <90 mmHg or diastolic blood pressure <50 mmHg), or hypertension (defined as systolic blood pressure >139 mmHg or diastolic blood pressure >89 mmHg).
8. Any history of clinically significant organ system (cardiovascular, neurological, hepatic, hematopoietic, renal, pulmonary, endocrine, or gastrointestinal) disorders or ongoing infectious diseases; or any other conditions that might interfere with the absorption, distribution, metabolism or excretion of the study drug, or that would place the subject at increased risk.
9. Use of marijuana (directly or indirectly) within 90 days prior to drug administration and during the course of the study.
10. History of treatment for alcohol abuse, significant mental illness, physical dependence to any opioid, barbiturates, amphetamines, cocaine, or benzodiazepines in the past 10 years.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2011-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Rate and extent of absorption | 48 hours
  The plasma concentration versus time data of dronabinol and its metabolite (11-hydroxy-delta-9-tetrahydrocannabinol) will be analyzed. The PK parameters Cmax, AUC0-t and AUCinf for delta-9-tetrahydrocannabinol will be calculated and used as the measures for comparative bioavailability assessment of dronabinol oral solution versus the innovator capsule product.

CONTACTS AND LOCATIONS:
Overall Officials: Joe Juren, M.D., Principal Investigator — Worldwide Clinical Trials
Locations (1):
- Worldwide Clinical Trials Drug Development Solutions, Austin, Texas, United States